CLINICAL TRIAL: NCT06304051
Title: Comparative Study of Effect of Intermittent Oral Enteral Nutrition Tube in Tracheostomized Patients With Intracerebral Hemorrhage
Brief Title: Effect of Intermittent Oral Enteral Nutrition Tube in Tracheostomized Patients With Intracerebral Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad (Other)
Responsible Party: Sponsor-Investigator, Muhammad, Research Director, Ahmadu Bello University Teaching Hospital
Organization: Ahmadu Bello University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Naochuxue-IOE
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Oro-esophageal Tube Feeding (Active Comparator): the nasogastric tube was removed, and Intermittent oro-esophageal tube feeding was initiated for nutrition support within 4 hours after completing the admission assessment, following the standard Intermittent oro-esophageal tube feeding procedure.
  Interventions: Device: Intermittent Oro-esophageal Tube Feeding
- Nasogastric Tube (Active Comparator): This group was provided with nutrition support by the indwelling nasogastric tube. The entire feeding process strictly followed the standardized procedure for nasogastric feeding.
  Interventions: Device: Nasogastric Tube Feeding

INTERVENTIONS:
Device: Intermittent Oro-esophageal Tube Feeding — Before each feeding, inside and outside of the tube was cleaned with water. During feeding, the patient should maintain a semi-reclining or sitting position with mouth opened, and the tube was inserted slowly and smoothly into the upper part of the esophagus by medical staffs while the appropriate depth of intubation was checked with the calibration markings on the tube wall. The distance from the incisors to the head part of the tube should be between 22-25 cm. However, the specific depth should be evaluated based on patients' feedback and adjusted accordingly. After insertion, the tail part of the tube should be put into a container full of water and the absence of continuous bubbles indicated a successful intubation. Then, the feeding was to be conducted three times per day with 50 ml per minute and 400-600ml for each feeding.
  Arms: Intermittent Oro-esophageal Tube Feeding
Device: Nasogastric Tube Feeding — Within 4 hours after admission, the placement of the feeding tube was conducted by professional medical staffs and after intubation, the tube was secured to the patient's cheek with medical tape. The feeding was conducted once every 3-4 hours, with 200-300ml each time. The total feeding volume was determined based on daily requirements. The feeding content was formulated by the nutritionists based on the patient's condition and relevant guidelines to reach the energy demand as 20-25 kcal/kg/day and protein supplementation of 1.2-2.0 g/kg/day for both two groups. For patients with limited tube feeding compliance, the investigators made appropriate adjustments to ensure that they were not at risk of severe malnutrition as much as possible.
  Arms: Nasogastric Tube

SUMMARY:
This was a multicenter, prospective, randomized controlled clinical trail involved tracheostomized patients with Intracerebral Hemorrhage.

The goal of this clinical trial is to compare the clinical effect of Intermittent Oro-esophageal Tube Feeding vs Nasogastric Tube Feeding in Tracheostomized Patients with Intracerebral Hemorrhage. The main questions it aims to answer are:

Compared to Nasogastric Tube Feeding, can the Intermittent Oro-esophageal Tube Feeding better improve the nutritional status, extubation of tracheostomy tube, pulmonary infection, neurological deficit of Patients with Intracerebral Hemorrhage Compared to Nasogastric Tube Feeding, is the Intermittent Oro-esophageal Tube Feeding safer.

Participants will be divided into two groups randomly, with different nutritional support respectively.

DETAILED DESCRIPTION:
Safe and efficient enteral nutrition support for tracheostomized patients with intracerebral hemorrhage continues to be a challenge.The goal of this clinical trial is to compare the clinical effect of Intermittent Oro-esophageal Tube Feeding vs Nasogastric Tube Feeding in Tracheostomized Patients with Intracerebral Hemorrhage. The main questions it aims to answer are:

Compared to Nasogastric Tube Feeding, can the Intermittent Oro-esophageal Tube Feeding better improve the nutritional status, extubation of tracheostomy tube, pulmonary infection, neurological deficit of Patients with Intracerebral Hemorrhage Compared to Nasogastric Tube Feeding, is the Intermittent Oro-esophageal Tube Feeding safer.

Participants will be divided into two groups randomly, with different nutritional support respectively.

ELIGIBILITY:
Inclusion Criteria:

* meeting the diagnostic criteria for Intracerebral Hemorrhage.
* with placement of a tracheotomy tube.
* requiring enteral nutrition support.
* age over 18 years.
* able to cooperate with treatment and questionnaire investigation.

Exclusion Criteria:

* combined with tumors in the head, neck, esophagus, or gastrointestinal tract
* an abnormal structure observed in the oral, pharyngeal, nasal regions or esophagus
* with unstable vital signs or severe dysfunction of organs including heart, liver, lungs, or kidneys
* with severe hemorrhagic disease or bleeding tendency;
* with dysphagia caused by non-stroke-related reasons in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Number of cases of successful extubation | day 30
  The Number of tracheostomized patients for both groups was recorded and compared. The parameters or criteria for extubation were: 1) stable clinical condition and a respiratory rate of 12-22 breaths per minute. 2) strong coughing ability and minimal airway secretions. 3) after completing a trial of tracheostomy tube capping, patients showed no fever, dyspnea, or asthma within 72 hours. Additionally, their blood oxygen saturation remained above 95% and normal oxygen partial pressure was observed

SECONDARY OUTCOMES:
Body mass index | day 1 and day 30
  Weight and height will be combined to report Body mass index in kg/m^2
Serum albumin level | day 1 and day 30
  Serum albumin was recorded via blood routine test.(Alb, g/L)
Hemoglobin level | day 1 and day 30
  Hemoglobin was recorded via blood routine test.(Hb, mg/L)
Clinical Pulmonary Infection Score | day 1 and day 30
  The Clinical Pulmonary Infection Score was recruited for evaluation, with specific assessment indicators such as body temperature, white blood cell count, respiratory secretions, chest X-rays, oxygenation index. The total scores ranged from 0 to 12, with a higher score indicated a more severe pulmonary infection

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Doctor, Study Chair — Site Coordinator of United Medical Group
Locations (2):
- China (2):
  - Fu shu afi. Hos., Huabei
  - Mingzhou Hos., Huaibei

IPD SHARING:
Plan to Share IPD: No